CLINICAL TRIAL: NCT05174494
Title: Impact of Non Surgical Periodontal Treatment on Serum NT-proBNP Levels
Brief Title: Impact of Periodontal Treatment on NT-proBNP Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, Dr., University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121/20/PO
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Periodontitis
Keywords: Periodontitis; serum markers; CRP; NT-proBNP
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Each selected patient underwent randomly, without anaesthesia, after recording periodontal parameters, the two following treatments: in one, maxillary quadrants were treated as conventional Scaling and Root Planing (SRP), while the control group undergo to standard oral hygiene treatment.
Who Masked: Participant, Investigator
Masking Description: Though sealed envelopes both clinicians and patients were masked to the selected treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full mouth non surgical periodontal treatment (Active Comparator): Each selected subject underwent to full mouth SRP.
  Interventions: Diagnostic Test: Evaluation of serum CRP and NT-proBNP
- Control (Placebo Comparator): Each selected subject underwent full mouth traditional oral hygiene.
  Interventions: Diagnostic Test: Evaluation of serum CRP and NT-proBNP

INTERVENTIONS:
Diagnostic Test: Evaluation of serum CRP and NT-proBNP — All patients were evaluated to 6-months post-treatment reduction of serum CRP and NT-proBNP

SUMMARY:
In light of the controversy that are already approved but that however still exists regarding the efficacy and influence the management of Periodontitis, the aim of this study was to evaluates, at 6-months follow-up, the post-treatment clinical and serum parameters in patients with periodontitis, treated by either Intensive scaling and root planing (SRP) treatment versus conventional oral hygiene treatment on serum CRP and NT-proBNP levels.

The null hypothesis to invalidate was that there were no variations, in relation to clinical and serum CRP and NT-proBNP.

DETAILED DESCRIPTION:
This trial was conducted in accordance with the World Medical Association's Declaration of Helsinki of 1975, and reviewed in 2016. The local ethical committee approved the study protocol and each patient was carefully informed about the possible inherent risks of the study and provided their informed written consent.

Subjects with a diagnosis of periodontitis were enrolled in this clinical trial. The inclusion criteria were: 1) good condition of general health, 2) a minimum of 2 teeth for each quadrant with a Pocket Depth (PD) ranging from 4-6 mm, 3) no involvement of the furcation, 4) a minimum of a six teeth per quadrant, respectively. The exclusion criteria were: 1) periodontal therapy during the last 12 months, 2) assumption of antibiotics during the last 6 months, 3) pregnancy, 4) any systemic condition which might affect the effects of the study treatment, 5) previous or current radiation or immunosuppressive therapies, 5) use of mouthwash containing antimicrobials during the previous 3 months, 6) no use of hormonal contraceptives, 7) medication by anti-inflammatory and immunosuppressive drugs, 8) previous history of hard-drinking, 9) smoking, 10) class II and III tooth mobility. Patients randomly undergo to full mouth SRP (test group) or oral hygiene treatment (control group)

ELIGIBILITY:
Inclusion Criteria:

* good condition of general health
* a minimum of 2 teeth for each quadrant with
* Pocket Depth (PD) ranging from 4-6 mm
* no involvement of the furcation
* a minimum of a six teeth per quadrant, respectively

Exclusion Criteria:

* periodontal therapy during the last 12 months
* assumption of antibiotics during the last 6 months
* pregnancy
* any systemic condition which might affect the effects of the study treatment
* previous or current radiation or immunosuppressive therapies
* use of mouthwash containing antimicrobials during the previous 3 months
* no use of hormonal contraceptives
* medication by anti-inflammatory and immunosuppressive drugs
* previous history of hard drinking
* smoking
* class II and III tooth mobility

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change of Clinical Attachment Level | 6-months
  Change of periodontal Clinical Attachment Level

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- University of Catania, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: Yes
Publish study results and IDP sharing plan
Supporting Information: Study Protocol
Time Frame: 1-year
Access Criteria: Pubmed
URL: https://pubmed.ncbi.nlm.nih.gov/